CLINICAL TRIAL: NCT00525616
Title: Assessment of Rituximab Efficiency and Tolerance in Treatment of Bullous Pemphigoid.
Brief Title: Efficiency and Tolerance of Rituximab (mabthéra) in Bullous Pemphigoid
Acronym: Rituximab2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006/101/HP
Record Dates: First submitted 2007-07-20; First posted 2007-09-06 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Bullous Pemphigoid
Keywords: bullous pemphigoid; mabthera
MeSH Terms: conditions — Pemphigoid, Bullous | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab (Experimental): Treatment consists of two slow intravenous infusions of rituximab 1000mg to 15 days apart with local corticosteroid .
  Interventions: Drug: Mabthera

INTERVENTIONS:
Drug: Mabthera — Two IV perfusions of 1000mg at 15 days intervals

SUMMARY:
The aim of the study is to assess that it will be possible to control with a single cycle of rituximab patient with bullous pemphigoid.

DETAILED DESCRIPTION:
The objective of this study is to assess the efficacy and tolerance of a single cycle of rituximab in control of bullous pemphigoid.

the main objects are :

1. to assess that a single cycle of rituximab is able to control patient with corticosteroid-dependent bullous pemphigoid,
2. to avoid the use of corticosteroid in long time,
3. to evaluate duration of control disease and side effect with a single cycle of rituximab.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 and < 80
* karnofsky >= 50%
* bullous pemphigoid clinical indication
* cortico-dependent bullous pemphigoid in relapse for the second time
* contraception used in female patient
* consent obtained from patient

Exclusion Criteria:

* localized bullous pemphigoid in relapse (<400cm2)
* pemphigoid of pregnancy
* dermatosis with IgA
* pemphigoid with mucous damage
* pregnant woman or nursing mother
* woman able to have a baby and without contraception during the clinical trial period
* age < 18 or > 80
* karnovsky < 50%
* significant disease or uncontrolled disease
* serious antecedents of allergy or anaphylactic reaction with human monoclonal antibody
* patient with depletion lymphocytic treatment or with initial rituximab treatment
* unstable angina or ischemic heart disease
* cardiac insufficiency
* cardiac rhythm trouble uncontrolled
* evolutive infection
* immunodepression
* neutrophil polynuclear in blood < 1.5 G/l and /or platelet blood concentration < 75G/l
* positive HIV serology
* positive hepatitis B and / or C serology
* concomitant immunodepressor treatment able to induce depletion lymphocytic treatment
* no consentment
* antecedent of serious chronic or recurrent infection or other underlying pathology able to induce serious infection
* antecedent of deep tissue infection occurred the previous year of inclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Clinical and biological controls of bullous pemphigoid were estimated every seven days during a period of 1 month and every month during a period of 2 years. | 2 years

SECONDARY OUTCOMES:
Adverse reactions will be estimated during all the period of this clinical trial | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Pascal JOLY, MD-PHD, Principal Investigator — Clinique Dermatologique - Hôpital Charles Nicolle
Locations (1):
- Rouen University Hospital, Direction de la Recherche et de l'Innovation,, Rouen, France